CLINICAL TRIAL: NCT00188630
Title: The PRIME (Perioperative Renal Insufficiency Management) Study: A Randomized, Double-blinded, Placebo-controlled Trial of N-acetylcysteine for Preventing Renal Injury After Cardiac Surgery.
Brief Title: N-Acetylcysteine for Preventing Renal Injury After Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Scott Beattie, Toronto General Hospital, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UHN REB 03-0376-B; HSFO5231
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Heart Disease; Acute Renal Failure
Keywords: Cardiac Surgery; Acute Renal Failure; N-acetylcysteine; Cardiopulmonary bypass
MeSH Terms: conditions — Heart Diseases; Acute Kidney Injury | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- N-Acetylcysteine (Active Comparator): IV NAC as a 100mg/kg bolus at the start of the surgical procedure (prior to the initiation of CPB), followed by a 10 mg/kg/hr infusion until 4 hours after completion of surgery
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): The control arm will instead receive placebo (5% dextrose solution), both as a bolus and infusion.
  Interventions: Other: 5% dextrose solution

INTERVENTIONS:
Drug: N-acetylcysteine
  Arms: N-Acetylcysteine
Other: 5% dextrose solution
  Arms: Placebo

SUMMARY:
Cardiac surgery improves the survival and quality of life of people with heart disease. Nonetheless, several complications continue to adversely affect outcomes following cardiac surgery. Kidney failure is a particularly important complication that is associated with increased death and duration of hospitalization. The most severe form of postoperative kidney failure, the need for dialysis, is uncommon at present. It is however likely to increase in the future. Patients undergoing cardiac surgery are getting older with more heart failure, diabetes, high blood pressure, and pre-existing kidney disease. Given that these are risk factors for postoperative kidney injury, dialysis rates will likely increase. Although multiple therapies have been tested, none have prevented postoperative kidney failure. N-acetylcysteine (NAC) is a drug that is commonly used to treat Tylenol overdoses. Over the past 2 years, it has also been used to prevent kidney damage after exposure to IV dye. There is good evidence that NAC will reduce kidney damage after IV dye exposure. There are strong reasons to believe that NAC may also prevent postoperative kidney failure. NAC is safe. Its major side-effects are allergic reactions, but serious reactions are rare. Since dialysis is uncommon, large studies are needed to determine if NAC prevents postoperative dialysis. In this situation, a pilot study is needed to determine if such a large trial is feasible. This proposal describes a pilot study. We will determine NAC's effects on creatinine clearance, a measure of how well the kidney works. Reduced creatinine clearance is closely related to dialysis and death after cardiac surgery. This biological marker allows us to determine NAC's effects on kidney function with a reduced sample size. If NAC improves creatinine clearance, it would suggest that NAC prevents postoperative dialysis, and would justify a larger study. A pilot study will help us estimate how many patients will be willing to participate in similar studies, vital for planning a future large study. Finally, our results will estimate how well NAC will reduce dialysis rates. This is needed for calculating the sample size for future studies.The study design is a randomized, double-blinded, placebo-controlled clinical trial among patients undergoing bypass surgery or heart valve surgery at the Toronto General Hospital (Toronto, ON). We will recruit 176 people who are at increased risk for developing kidney failure after surgery. Participants will receive either NAC or sugar solution during their operation. If participants have returned home within a month of surgery, they will be contacted at home on the 30th day after surgery to determine if they had any kidney-related problems since returning home. All participants will return to the Toronto General Hospital (TGH) during the 8th week after surgery for creatinine blood test and weight.

ELIGIBILITY:
Inclusion Criteria:

* CABG surgery under cardiopulmonary bypass AND/OR Valve replacement/repair surgery under cardiopulmonary bypass
* Preoperative creatinine clearance (Cockcroft-Gault equation) <= 60 mL/min.
* Age above 18 years
* Informed consent

Exclusion Criteria:

* Preoperative need for renal replacement therapy
* Preoperative serum creatinine concentration >= 300 mmol/L
* Prior adverse reaction to NAC with significant systemic symptoms (generalized rash, urticaria, bronchospasm, hypotension)
* Preoperative intra-aortic balloon pump support and/or inotropes/vasopressors
* Recent coronary angiography or intravenous dye exposure (<= 24 hours) preceding surgery
* Planned intraoperative deep hypothermic circulatory arrest
* Pregnancy
* Chronic hepatitis or hepatic cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2003-07; Primary Completion 2007-02 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Maximum percent decline in calculated creatinine clearance (Cockcroft-Gault formula) in first 72 hours following surgery. | 72 hours following surgery

SECONDARY OUTCOMES:
Maximum increase in serum creatinine concentration over first 72 hours following surgery. | 72 hours following surgery
Increase in serum creatinine >= 0.5 mg/dL from baseline over first 72 hours following surgery (dichotomous outcome). | 72 hours following surgery
Maximum percent decline in calculated creatinine clearance (Cockcroft-Gault formula) >= 25% in first 72 hours following surgery (dichotomous outcome). | 72 hours following surgery
Percent change in calculated creatinine clearance (Cockcroft-Gault formula) at hospital discharge. | hospital discharge
Maximum percent decline in calculated creatinine clearance (Cockcroft-Gault formula) at 8 weeks following surgery. | 8 weeks followiing surgery
30-day need for renal replacement therapy | 30 day inclusive
30-day all-cause mortality | 30 day follow up
Length of stay in intensive care unit (postoperative) | Duration of stay in the ICU
Length of stay in hospital (postoperative) | Until discharge form hospital
24-hour fluid perioperative fluid balance | 24 hours
24-hour urine output | 24 hour
Adverse perioperative event | Intra operative measure

CONTACTS AND LOCATIONS:
Overall Officials: William S Beattie, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (1):
- Toronto General Hospital, UHN, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Wijeysundera DN, Karkouti K, Rao V, Granton JT, Chan CT, Raban R, Carroll J, Poonawala H, Beattie WS. N-acetylcysteine is associated with increased blood loss and blood product utilization during cardiac surgery. Crit Care Med. 2009 Jun;37(6):1929-34. doi: 10.1097/CCM.0b013e31819ffed4. PMID 19384218